CLINICAL TRIAL: NCT02437461
Title: Dosing of Intra-articular Triamcinolone Hexacetonide for Knee Synovitis in Chronic Polyarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Thomas Weitoft, MD, PhD, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TW77
Record Dates: First submitted 2015-04-30; First posted 2015-05-07 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Arthritis of the Knee
Keywords: knee synovitis; triamcinolone hexacetonide; treatment response
MeSH Terms: interventions — triamcinolone hexacetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single dose 20 mg (Active Comparator): Intraarticular injection of triamcinolone hexacetonide
  Interventions: Drug: Triamcinolone hexacetonide
- single dose 40 mg (Experimental): Intraarticular injection of triamcinolone hexacetonide
  Interventions: Drug: Triamcinolone hexacetonide

INTERVENTIONS:
Drug: Triamcinolone hexacetonide — intraarticular knee injection
  Other Names: Lederspan

SUMMARY:
This prospective randomised controlled single blind trial comparing the relapse rate in 6 months for 20 mg versus 40 mg intraarticular triamcinolone hexacetonide (Lederspan®) for knee synovitis in patients with rheumatoid arthritis (RA) and psoriatic artritis (PsoA) is performed to find the optimal dose to use.

DETAILED DESCRIPTION:
Background:

Triamcinolone hecacetonide (THA) has been used for local intraarticular injecton treatment for knee synovitis in decades, but no dose finding studies have been performed. In the literature the doses for knee injections vary between 20 mg and 80 mg, depending on local traditions.

The aim of the present study is to find the optimal THA dosing, comparing the relapse rate during a 6 month observation period for the two most used dosages .

Methods:

Adult patients with RA or PsoA with treatment demands for ongoing knee synovitis are recruited at the Rheumatology Departments in Gävle and Falun. After informed consent patient characteristics,(age, sex, medical treatment), clinical and laboratory parameters of disease activity (DAS28, CRP), as well as degree of functional impairment (HAQ) are collected. A radiographic examination of the knee is performed and assessed (using Larsen Dale index) by an independent radiologist. The patients are allocated to either 20 mg or 40 mg THA using the randomisation dose which is hidden in prepared closed envelopes. After complete synovial fluid aspiration the THA dose is injected . The patients are told to contact the rheumatology department if no treatment response or if symtoms from the treated knee recurr. If so, the knee is examined again and if synovitis is confirmed a relapse is registered. Time from injection to relapse is calculated. Patients without relapse are called after 6 months to confirm they still are well and that no unknown relapse have occurred. When the observation period for the last included patient is finished the relapse rate between the 20 mg THA group is compared with the 40 mg THA Group.

ELIGIBILITY:
Inclusion Criteria: synovitis of the knee, rheumatoid arthritis or psoriatic arthrthritis, written informed consent

-

Exclusion Criteria:

* inability to understand study information, function class 4 according to Steinbrocker, planning knee surgery, , joint infection, intraarticular glucocorticoid injection in this joint the past 3 months, oral glucocortoid treatment corresponding to >10 mg prednisolone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-06-20 (Estimated)

PRIMARY OUTCOMES:
arthritis relapse | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Weitoft, MD, PhD, Principal Investigator — Center for Research and Development Uppsala University/Region Gavleborg
Locations (1):
- Section of Rheumatology, Gävle hospital, Gävle, Sweden

REFERENCES:
- [Background] Weitoft T, Uddenfeldt P. Importance of synovial fluid aspiration when injecting intra-articular corticosteroids. Ann Rheum Dis. 2000 Mar;59(3):233-5. doi: 10.1136/ard.59.3.233. PMID 10700435
- [Background] Lopes RV, Furtado RN, Parmigiani L, Rosenfeld A, Fernandes AR, Natour J. Accuracy of intra-articular injections in peripheral joints performed blindly in patients with rheumatoid arthritis. Rheumatology (Oxford). 2008 Dec;47(12):1792-4. doi: 10.1093/rheumatology/ken355. Epub 2008 Sep 27. PMID 18820311
- [Background] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570
- [Background] Ekdahl C, Eberhardt K, Andersson SI, Svensson B. Assessing disability in patients with rheumatoid arthritis. Use of a Swedish version of the Stanford Health Assessment Questionnaire. Scand J Rheumatol. 1988;17(4):263-71. doi: 10.3109/03009748809098795. PMID 3187457
- [Background] Weitoft T, Ronnelid J, Knight A, Lysholm J, Saxne T, Larsson A. Outcome predictors of intra-articular glucocorticoid treatment for knee synovitis in patients with rheumatoid arthritis - a prospective cohort study. Arthritis Res Ther. 2014 Jun 20;16(3):R129. doi: 10.1186/ar4586. PMID 24950951
- [Background] Larsen A, Dale K. Standardized radiological examination of rheumatoid arthritis in therapeutical trials. In Dumonde DC, Jasani MK, eds. The recognition of antirheumatic drugs. Lancaster: MTP Press, 1978: 285-292
- [Background] Arnett FC, Edworthy SM, Bloch DA, McShane DJ, Fries JF, Cooper NS, Healey LA, Kaplan SR, Liang MH, Luthra HS, et al. The American Rheumatism Association 1987 revised criteria for the classification of rheumatoid arthritis. Arthritis Rheum. 1988 Mar;31(3):315-24. doi: 10.1002/art.1780310302. PMID 3358796
- [Background] Taylor W, Gladman D, Helliwell P, Marchesoni A, Mease P, Mielants H; CASPAR Study Group. Classification criteria for psoriatic arthritis: development of new criteria from a large international study. Arthritis Rheum. 2006 Aug;54(8):2665-73. doi: 10.1002/art.21972. PMID 16871531
- [Background] STEINBROCKER O, TRAEGER CH, BATTERMAN RC. Therapeutic criteria in rheumatoid arthritis. J Am Med Assoc. 1949 Jun 25;140(8):659-62. doi: 10.1001/jama.1949.02900430001001. No abstract available. PMID 18150288
- [Derived] Weitoft T, Oberg K. Dosing of intra-articular triamcinolone hexacetonide for knee synovitis in chronic polyarthritis: a randomized controlled study. Scand J Rheumatol. 2019 Jul;48(4):279-283. doi: 10.1080/03009742.2019.1571222. Epub 2019 Mar 7. PMID 30843453